CLINICAL TRIAL: NCT06387433
Title: Assessing the Effectiveness of an mHealth Intervention Versus the Usual Standard of Care for Improving Medication Adherence and Self-management Among Type II Diabetics in Pakistan: A Randomized Controlled Trial
Brief Title: Effectiveness of an mHealth Mobile App
Acronym: mHealth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Maria Atif, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mHealth; SG-222/R3-05/RDC/DUHS/1478 (Other Grant/Funding Number: National Institutes of Health Pakistan)
Record Dates: First submitted 2024-04-15; First posted 2024-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Type II Diabetes
Keywords: diabetes mellitus; mobile applications; Pakistan
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile app users (Experimental)
  Interventions: Behavioral: mobile app use
- mobile app non-users (No Intervention)

INTERVENTIONS:
Behavioral: mobile app use — The experimental group will use the mobile application while controlled group will not use mobile application. Investigators will assess the effectiveness of mobile application in ensuring medication adherence and self-management among diabetics in Pakistan
  Arms: mobile app users

SUMMARY:
Type II diabetes is a serious challenge for Pakistan. Not using medications properly increases healthcare costs and diabetes-related deaths. A mobile app in local language can improve medication adherence and self-management among diabetics. Therefore, in this 18 months long study researchers will develop a diabetes-related mobile application in Urdu, and will conduct a trial to assess whether it improves medication compliance and self-management, and how much economical this app would be compared to the usual standard of care for type II diabetics in Pakistan. This trial will be conducted at the National Institute of Diabetes and Endocrinology Karachi. The study participants will be divided in two groups. Only one group will use this application. Researchers will measure medication compliance and self-management through diabetes-specific blood test and self-reporting questionnaires between two groups. Researchers will also determine how much economic costs would be saved by using this app to improve medication compliance

DETAILED DESCRIPTION:
Type II diabetes continues to be a challenge for the resource-constrained healthcare system in Pakistan. Non-adherence to medications increases healthcare costs and disease-related mortality. Mobile health (mHealth), especially in local language, can improve medication adherence and self-management among diabetics. However, there are currently no validated diabetes-related apps available in Urdu for Pakistani population The objective of this study is to develop an android-compatible mobile application in Urdu, to assess its effectiveness in improving medication adherence and self-management, and to conduct an economic evaluation of this app against the usual standard of care for type II diabetics in Pakistan. This 18 months long randomized controlled trial will be conducted at the National Institute of Diabetes and Endocrinology Karachi. This bi-phasic study will involve the development and pilot testing of an android-compatible app, followed by an RCT to assess the effectiveness of this mobile app in improving medication adherence and self-management among type II diabetics in Pakistan. Medication adherence will be measured by the HbA1c levels and self-reported Morisky Medication Adherence Scale (Urdu version), while self- management will be assessed by Diabetes Self-Management Questionnaire (Urdu version). All outcomes will be assessed at 3 and 6 months. Intervention usability will be evaluated by the Mobile App Rating Scale (MARS) and economic effectiveness will be evaluated by EQ-5D-3L (Urdu version) to measure Quality Adjusted Life Years.

The expected outcome is the production of scientific evidence for the effectiveness and economic viability of a locally-validated mobile application for diabetes care and management in Pakistan

ELIGIBILITY:
Inclusion Criteria:

* Adults
* HbA1c more than or equal to 8.0 on most recent lab report within last 3 months
* able to comprehend Urdu language

Exclusion Criteria:

* type I diabetics,
* patients on continuous glucose monitoring,
* patients with severe mental or physical impairment,
* pregnant
* do not have access to smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
adherence to medication | baseline, 3 and 6 months
  measured by Morisky Medication Adherence Scale .For Morisky Medication Adherence Scale, a score of less than 6 will be considered low adherence and higher scores will indicate better adherence
self-management among diabetics | baseline, 3 and 6 months
  measured by Diabetes self-management questionnaire. This questionnaire has a scale from 0 to 10, with the score of 10 indicating the most effective self-care behaviour.
effective management of diabetes | baseline, 3 and 6 months
  Adherence to treatment will also be assessed by the HbA1c levelsHbA1c levels of 8% or more will be considered diabetic, with higher score indicating poor control of diabetes

SECONDARY OUTCOMES:
Intervention usability | measured at 6 months following intervention
  measured through Mobile Application Rating Scale. In this scale all points are rated on 5 point scale from 1 indicating 'inadequate' and 5 indicating 'excellent'
economic effectiveness of the app | measured at 6 months following intervention
  measured through EQ-5D-3L. calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Atif, Principal Investigator — Dow University of Health Sciences
Locations (1):
- National Institute of Diabetes and Endocrinology, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No